CLINICAL TRIAL: NCT02730078
Title: The Effectiveness of a Value-based Emotion-focused Educational Programme to Reduce Diabetes-related Distress in Malay Adults With Type 2 Diabetes (VEMOFIT): a Cluster Randomised Controlled Trial
Brief Title: Value-based Emotion-focused Educational Programme to Reduce Diabetes-related Distress
Acronym: VEMOFIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Collaborators: Ministry of Health, Malaysia (Other Government); UMC Utrecht (Other)
Responsible Party: Principal Investigator, Boon-How Chew, Associate Professor, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMRR- 15-1144-24803
Record Dates: First submitted 2016-03-29; First posted 2016-04-06 (Estimated); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Mood Disorders; Self Care; Primary Care
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Mood Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Attention-meetings (AG) (Active Comparator): Attention-control
  Interventions: Behavioral: Attention-meetings (AG)
- VEMOFIT (VG) (Experimental): Personal value exploration, disease education, emotional skills and goal setting.
  Interventions: Behavioral: VEMOFIT

INTERVENTIONS:
Behavioral: VEMOFIT — The VEMOFIT intervention involves four biweekly two hours sessions over a period of about six weeks, and a booster at three months follow-up. It consists of a mixture of 1) exploring illness perceptions and personal meanings of diabetes, 2) cognition-focused education on diabetes and practical skills in self-management and 3) emotion-focused training on recognising emotions in the self and others. Each group will consist of 10 to 12 participants of equal representation by the patients and their significant others.
  Other Names: Value-based emotion-focused educational programme
  Arms: VEMOFIT (VG)
Behavioral: Attention-meetings (AG) — Patients in the health clinics randomised to the AG, will receive the usual T2D care by the clinic doctors and education by the clinic paramedics based on the recommendations in the Malaysian clinical guidelines. At T1, T2 and T4, patients (not including their significant others) in AG will be gathered in groups of 10-12 people for the primary and secondary outcomes evaluation. This session will include general discussion on feeling about and coping with T2D, social support at home and satisfaction with treatment and care received at the respective clinics.
  Arms: Attention-meetings (AG)

SUMMARY:
The purpose of the clinical trial is to evaluate the effectiveness of a relatively simple and short value-based emotion-focused educational programme in adults with type 2 diabetes (VEMOFIT) on diabetes-related distress, depressive symptoms, illness perception, medication adherence, quality of life, diabetes self-efficacy, self-care and clinical outcomes.

DETAILED DESCRIPTION:
Type 2 diabetes (T2D) patients experience many psychosocial problems related to their diabetes, as well as social- and work-related relationships. These often lead to emotional disorders such as distress, stress, anxiety and depression. Without proper care, these patients use more often negative coping strategies and more frequently expect that their diabetes will negatively affect their future. A cluster randomised controlled trial will be conducted in 10 public health clinics (HC) in Malaysia. These clusters are eligible if they are providing standard diabetes care according to national clinical practice guidelines, not involved in similar trial and having nurses to be trained to deliver the VEMOFIT educational programmes. Pre-stratification by cluster size and geographic areas of the HCs will get randomised five HCs to the VEMOFIT group (VG) and attention-meetings group (AG), respectively.

ELIGIBILITY:
Inclusion Criteria:

* Malay patients
* Diagnosed with T2D for at least two years
* On regular follow-up with at least three visits in the past one year
* Have diabetes-related distress (mean DDS-17 score ≥ 3)
* Showing poor disease control (not reaching targets for one of the three biomarkers, namely HbA1c ≥ 8%, blood pressure ≥ 140/90 mmHg and LDL-C > 2.6 mmol/L)

Exclusion Criteria:

* Patients who are enrolled in other clinical studies
* Pregnant or lactating
* Having psychiatric/ psychological disorders that could impair judgments and memory
* Patients who cannot read or understand English or Malay
* Patients who scored ≥ 20 on the Patient Health Questionnaire-9 (PHQ-9) that suggest a severe depression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Diabetes-related distress | 6-week (immediate post-intervention) [T1]
  Measured with the 17-item Diabetes Distress Scale (DDS-17)
Diabetes-related distress | 6-month [T2]
  Measured with the 17-item Diabetes Distress Scale (DDS-17)
Diabetes-related distress | 12-month [T3]
  Measured with the 17-item Diabetes Distress Scale (DDS-17)

SECONDARY OUTCOMES:
Depression | 6-week (immediate post-intervention) [T1]
  Measured with the Patient Health Questionnaire (PHQ-9)
Depression | 6-month [T2]
  Measured with the Patient Health Questionnaire (PHQ-9)
Depression | 12-month [T3]
  Measured with the Patient Health Questionnaire (PHQ-9)
Illness perception | 6-week (immediate post-intervention) [T1]
  Measured with the Brief Illness Perception Questionnaire (BIPQ)
Illness perception | 6-month [T2]
  Measured with the Brief Illness Perception Questionnaire (BIPQ)
Illness perception | 12-month [T3]
  Measured with the Brief Illness Perception Questionnaire (BIPQ)
Quality of life | 6-month [T2]
  Measured with the WHOQOL-BREF
Quality of life | 12-month [T3]
  Measured with the WHOQOL-BREF
Self-efficacy | 6-week (immediate post-intervention) [T1]
  Measured by the Diabetes Management Self Efficacy Scale (DMSES)
Self-efficacy | 6-month [T2]
  Measured by the Diabetes Management Self Efficacy Scale (DMSES)
Self-efficacy | 12-month [T3]
  Measured by the Diabetes Management Self Efficacy Scale (DMSES)
Self-care behaviours | 6-week (immediate post-intervention) [T1]
  Measured with the Diabetes Self-Care Activities (SDSCA) scale
Self-care behaviours | 6-month [T2]
  Measured with the Diabetes Self-Care Activities (SDSCA) scale
Self-care behaviours | 12-month [T3]
  Measured with the Diabetes Self-Care Activities (SDSCA) scale
Positive emotions | 6-week (immediate post-intervention) [T1]
  Measure by the Positive Affects subscale of the Center for Epidemiologic Studies Depression Scale (PA-CESD)
Positive emotions | 6-month [T2]
  Measure by the Positive Affects subscale of the Center for Epidemiologic Studies Depression Scale (PA-CESD)
Positive emotions | 12-month [T3]
  Measure by the Positive Affects subscale of the Center for Epidemiologic Studies Depression Scale (PA-CESD)
HbA1c | 6-week (immediate post-intervention) [T1]
HbA1c | 6-month [T2]
HbA1c | 12-month [T3]
Blood pressure | 6-week (immediate post-intervention) [T1]
  systolic and diastolic blood pressure
Blood Pressure | 6-month [T2]
  systolic and diastolic blood pressure
Blood pressure | 12-month [T3]
  systolic and diastolic blood pressure
LDL-cholesterol | 6-week (immediate post-intervention) [T1]
  lipid profiles
LDL-cholesterol | 6-month [T2]
  lipid profiles
LDL-cholesterol | 12-month [T3]
  lipid profiles

OTHER OUTCOMES:
Health-care utilisation/hospitalisation | 6-month [T2]
  Number of visits to healthcare facilities including hospitalisation, patient's record and diary used in the study
Health-care utilisation/hospitalisation | 12-month [T3]
  Number of visits to healthcare facilities including hospitalisation, patient's record and diary used in the study
Adverse event | 6-week (immediate post-intervention) [T1]
  Number of hypoglycaemia and extreme negative emotions as recorded in participant's diary
Adverse event | 6-month [T2]
  Number of hypoglycaemia and extreme negative emotions as recorded in participant's diary
Adverse event | 12-month [T3]
  Number of hypoglycaemia and extreme negative emotions as recorded in participant's diary

CONTACTS AND LOCATIONS:
Overall Officials: Boon-How Chew, MMed, Principal Investigator — Universiti Putra Malaysia

IPD SHARING:
Plan to Share IPD: Yes
Anonymous data will be accessible publicly via the figshare.

REFERENCES:
- [Background] Chew BH, Vos RC, Shariff Ghazali S, Shamsuddin NH, Fernandez A, Mukhtar F, Ismail M, Mohd Ahad A, Sundram NN, Ali SZ, Rutten GE. The effectiveness of a value-based EMOtion-cognition-Focused educatIonal programme to reduce diabetes-related distress in Malay adults with Type 2 diabetes (VEMOFIT): study protocol for a cluster randomised controlled trial. BMC Endocr Disord. 2017 Apr 4;17(1):22. doi: 10.1186/s12902-017-0172-8. PMID 28376921
- [Background] Chew BH, Vos RC, Metzendorf MI, Scholten RJ, Rutten GE. Psychological interventions for diabetes-related distress in adults with type 2 diabetes mellitus. Cochrane Database Syst Rev. 2017 Sep 27;9(9):CD011469. doi: 10.1002/14651858.CD011469.pub2. PMID 28954185
- [Background] Chew BH, Fernandez A, Shariff-Ghazali S. Psychological interventions for behavioral adjustments in diabetes care - a value-based approach to disease control. Psychol Res Behav Manag. 2018 May 4;11:145-155. doi: 10.2147/PRBM.S117224. eCollection 2018. PMID 29765258
- [Background] Chew BH, Shariff-Ghazali S, Fernandez A. Psychological aspects of diabetes care: Effecting behavioral change in patients. World J Diabetes. 2014 Dec 15;5(6):796-808. doi: 10.4239/wjd.v5.i6.796. PMID 25512782
- [Background] Chew BH, Mukhtar F, Sherina MS, Paimin F, Hassan NH, Jamaludin NK. The reliability and validity of the Malay version 17-item Diabetes Distress Scale. Malays Fam Physician. 2015 Aug 31;10(2):22-35. eCollection 2015. PMID 27099658
- [Result] Chew BH, Vos RC, Stellato RK, Ismail M, Rutten GEHM. The effectiveness of an emotion-focused educational programme in reducing diabetes distress in adults with Type 2 diabetes mellitus (VEMOFIT): a cluster randomized controlled trial. Diabet Med. 2018 Jun;35(6):750-759. doi: 10.1111/dme.13615. Epub 2018 Mar 30. PMID 29505098
- [Result] Chew BH, Vos RC, Fernandez A, Shariff Ghazali S, Shamsuddin NH, Ismail M, Rutten GEHM. The effectiveness of an emotion-focused educational programme in reducing diabetes distress in adults with type 2 diabetes mellitus at 12-month follow-up: a cluster randomized controlled trial. Ther Adv Endocrinol Metab. 2019 May 31;10:2042018819853761. doi: 10.1177/2042018819853761. eCollection 2019. PMID 31210922
- [Derived] Chew BH, Vos RC, Heijmans M, Shariff-Ghazali S, Fernandez A, Rutten GEHM. Validity and reliability of a Malay version of the brief illness perception questionnaire for patients with type 2 diabetes mellitus. BMC Med Res Methodol. 2017 Aug 3;17(1):118. doi: 10.1186/s12874-017-0394-5. PMID 28774271
- See also: Study protocol published in Springer BMC Endocrine Disorders — http://rdcu.be/qEPS